CLINICAL TRIAL: NCT01117116
Title: Sub-Sensitivity to Long-Acting Bronchodilators (LABA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GSK LABA
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination; Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fluticasone propionate and salmeterol (Active Comparator)
  Interventions: Drug: fluticasone propionate and salmeterol; Drug: budesonide and formoterol
- budesonide and formoterol (Active Comparator)
  Interventions: Drug: fluticasone propionate and salmeterol; Drug: budesonide and formoterol

INTERVENTIONS:
Drug: fluticasone propionate and salmeterol — 45/4.5 two puffs twice daily
  Other Names: Advair
Drug: budesonide and formoterol — 80/4.5 two puffs twice daily
  Other Names: Symbicort

SUMMARY:
The purpose of this study is to look at whether Advair® and SYMBICORT® have different effects on airway constriction by means of methacholine challenge testing.

ELIGIBILITY:
Inclusion Criteria:

* 20 subjects males or females 18-65 years of age with physician diagnosed asthma Diagnosis of asthma > 12 months Currently on 2 puffs SABA bid. Baseline percent FEV1 of greater than 60% and less than or equal to 100% 12% reversibility in the previous 12 months 12% reversibility at Screening Visit Positive MTC (≤ 8mg/ml) at the end of 2 week Run-In Currently symptomatic with ACT score less than 19 at the end of run in on ICS ≥ 200 and ≤ 400 ug/day Non-smoker or ex-smoker with < 10 pk year who stopped > 1 year ago

Exclusion Criteria:

* Asthma exacerbation, significant airflow obstruction, or respiratory infection between Visits 0 and 2. Patients who fail screening because of one of these events may be re-screened once (at least 4 weeks after recovery from the event).

Pre-existing lung disease other than asthma, including active infections Clinically significant medical disease that is uncontrolled despite treatment or is likely in the opinion of the investigator to require a change in therapy during the study Noncompliance or inability to participate in all assessments. Current smoker or former smoker with a lifetime smoking history of ≥ 10 pack-years. A current smoker is defined as someone who has smoked one or more cigarettes per day (or marijuana or a pipe or cigar) for >/= 30 days within the 24 months prior to Visit 1.

Any individual who smokes (cigarettes, marijuana, pipe, or cigar) occasionally, even if for < 30 days in the 24 months Prior to Visit 1, must agree to abstain from all smoking from the time of consent through completion.

History of substance abuse that may impair or risk the patient's full participation in the study, in the judgment of the investigator.

Participation in another interventional clinical trial (including a trial of an approved drug or an interventional study that does not include medication) within 30 days or 5 half-lives of the investigational agent, whichever is longer.

Women with a positive urine pregnancy test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Improvement in PC20 | Study Completion
  Improvements in PC20 as measured by methacholine challenge between the two treatment groups at the end of the first 4 week period to determine efficacy between low dose Advair and Symbicort.

SECONDARY OUTCOMES:
Changes in FEV1 | Study Completion
  Changes in peak pre-bronchodilator FEV1 [measured at hours 10, 11, 12 post evening dose] over the four week treatment periods and over each 12 hour dosing period (pre evening dose FEV1).

CONTACTS AND LOCATIONS:
Overall Officials: Rohit K Katial, M.D., Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States